CLINICAL TRIAL: NCT05580679
Title: The Effect of Abdominal Massage on Managing Constipation in Palliative Care Patients
Brief Title: Effect of Abdominal Massage on Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Özge Uçar, Research Assistant, Bartın Unıversity
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1919B012101971
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Constipation; Abdominal Pain; Palliative Care
Keywords: palliative; palliative care; nursing; abdominal massage; constipation
MeSH Terms: conditions — Constipation; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trials
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal massage group (Experimental): Abdominal massage using for evaluation of constipation.
  Interventions: Other: Abdominal massage
- Standart care group (No Intervention): No intervention palliative care patient

INTERVENTIONS:
Other: Abdominal massage — Application time of the massage: 30 minutes after meals, twice a day, at 10:00 in the morning and at 16:00 in the evening.
  Application time of the massage: 15 minutes each Materials needed: Gloves, Liquid Vaseline, Paper Towel Massage methods used: Efflorage, Petrissage, Vibration
  Arms: Abdominal massage group

SUMMARY:
Constipation is defined as infrequent defecation or difficulty in evacuation. Although the constipation problem is mostly self-managed by the patients, 22% mostly refer to primary health care providers (>50%), resulting in large expenditures for diagnostic tests and treatments. According to studies conducted in our country, the incidence of constipation varies between 22-40%, while it is stated that the prevalence of constipation in hospitalized patients is 79%. Annual medical costs due to constipation are estimated to exceed 230 million dollars. Pharmacological and non-pharmacological methods are used in the management of constipation, which is one of the most common symptoms in the hospital. The use of non-pharmacological methods is recommended due to the possibility of side effects and cost of pharmacological methods. However, the prevalence of use of non-pharmacological methods in the clinic is low. Nurses need to have knowledge about non-pharmacological methods in order to manage the problem of constipation, which is one of the most common symptoms in the hospital. Abdominal massage, which is included in the Nursing Interventions Classification (NIC), is an application performed with manipulations such as pressure and rubbing on certain points on the body to reduce pain, provide relaxation and relaxation, prevent and reduce nausea, and prevent constipation.

DETAILED DESCRIPTION:
Introduction: Constipation is defined as infrequent defecation or difficulty in evacuation. Although the constipation problem is mostly self-managed by the patients, 22% mostly refer to primary health care providers (>50%), resulting in large expenditures for diagnostic tests and treatments. According to studies conducted in our country, the incidence of constipation varies between 22-40%, while it is stated that the prevalence of constipation in hospitalized patients is 79%. Annual medical costs due to constipation are estimated to exceed 230 million dollars. Pharmacological and non-pharmacological methods are used in the management of constipation, which is one of the most common symptoms in the hospital. The use of non-pharmacological methods is recommended due to the possibility of side effects and cost of pharmacological methods. However, the prevalence of use of non-pharmacological methods in the clinic is low. Nurses need to have knowledge about non-pharmacological methods in order to manage the problem of constipation, which is one of the most common symptoms in the hospital. Abdominal massage, which is included in the Nursing Interventions Classification (NIC), is an application performed with manipulations such as pressure and rubbing on certain points on the body to reduce pain, provide relaxation and relaxation, prevent and reduce nausea, and prevent constipation.

Objective: This study was planned to examine the effect of abdominal massage on the management of constipation in palliative care patients.

Method: The project will be carried out in a state hospital in Bartın, between 01.09.2021 and 01.09.2022, in the palliative care service, with patients over 18 years of age, without a history of gastrointestinal cancer, history of abdominal surgery or abdominal hernia, and hospitalized for at least 7 days. Palliative care patients hospitalized in Bartın State Hospital in the last 1 year will form the universe. Sample calculation will be made with G power analysis and the participants will be divided into experimental and control groups with block randomization. The patients in the experimental group will be given abdominal massage in the morning and evening every day for 1 week and the defecation status of the patients will be compared. The data will be recorded in the data collection form prepared in line with the literature. The data will be used in the patient identification form, Gastrointestinal Symptom Rating Scale, Constipation Evaluation Scale, Bristol Stool Consistency Scale. The collected data will be evaluated using the SPSS program.

Conclusion: With this project, the incidence of constipation in palliative patients will be determined and the knowledge and skills of nursing students on how to apply abdominal massage, which is one of the nursing practices, will increase. With their practice in this study, they will play an active role in the management of constipation in palliative patients, and they will be able to perform this practice in patients in various services throughout their education and professional lives.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering
* Being over 18 years old
* No history of gastrointestinal cancer, history of abdominal surgery or abdominal hernia
* At least 7 days of clinical treatment

Exclusion Criteria:

* Patient information form
* Gastrointestinal system rating scale
* Constipation assessment scale
* Bristol stool consistency scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
First measurements of defecation type. | 1-7 days
  First measurements of both group before intervention using by Bristol Stool Consistency Scale. The Bristol Stool Consistency Scale, developed by a team of gastroenterologists at the University of Bristol, UK; It is used to evaluate stool form and to have information about changes in bowel habits and a pathological formation that may occur in the intestine. This scale was designed to classify an individual's bowel movements in seven distinct categories of stool. According to the Bristol Stool Consistency Scale, Type 1 and Type 2 are constipation, Type 3 and Type 4 are normal stools, and Type 5, Type 6 and Type 7 are diarrhea. It is accepted that there is a direct relationship between stool shape and length of stay in the colon (Lewis and Heaton 1997).
First measurements of gastrointestinal symptoms | 1-7 days
  First measurements of both groups before the intervention using a Gastrointestinal Symptom Rating Scale.The Turkish validity and reliability of the scale, which was developed by Revicki et al. in 1998 to evaluate the symptoms frequently seen in gastrointestinal system disorders, was performed by Turan and Aştı in 2011. GSRS; It is a 15-item Likert-type scale with options starting from "no discomfort" to "very severe discomfort". Based on factor analysis, 15 items of the GSRS have five sub-dimensions: Abdominal Pain, Reflux, Diarrhea, Indigestion and Constipation. In the GSRS, how the individual felt in terms of gastrointestinal problems in the last week is questioned. High scores on the GSRS indicate that the symptoms are more severe (Revicki et al. 1998; Kaya and Turan 2011; Turan and Aştı 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Özge Uçar, Principal Investigator — Bartin University Health Science Faculty; Nursena Eren, Study Director — Bartin University Health Science Faculty; Nisa Ün, Study Chair — Bartin University Health Science Faculty; Erdem Altuner, Study Chair — Bartin University Health Science Faculty; İrem Yılmaz, Study Chair — Bartin University Health Science Faculty
Locations (1):
- Özge Uçar, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No